CLINICAL TRIAL: NCT02538055
Title: Using CERS to Optimize Quality of Life for Persons With Diabetes and Chronic Pain
Acronym: Living Healthy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Monika M. Safford, Professor, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R18HS019239 (AHRQ)
Record Dates: First submitted 2015-07-06; First posted 2015-09-02 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus; Chronic Pain
Keywords: Community Health Workers; Diabetes Mellitus; Chronic Pain
MeSH Terms: conditions — Diabetes Mellitus; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Health Program (Placebo Comparator): Participants in this arm worked with a Community Health Worker (CHW) who provided a general health program that consisted of didactic information of unrelated general health information. Participants received the same number of contacts with their CHW as the intervention arm. Participants and CHW interacted by telephone 8 times over 3 months.
  Interventions: Behavioral: General Health Program
- Living Healthy Program (Experimental): Participants in this arm worked with a Community Health Worker (CHW) who provided the Living Healthy Program. The Living Healthy Program was a cognitive-behavioral therapy based lifestyle modification program. Participants and CHW interacted by telephone 8 times over 3 months.
  Interventions: Behavioral: Living Healthy

INTERVENTIONS:
Behavioral: Living Healthy — This intervention tested the effects of a community health worker delivered lifestyle modification program based on cognitive behavioral therapy on diabetes and pain outcomes in individuals with diabetes and chronic pain.
  Arms: Living Healthy Program
Behavioral: General Health Program — Participants in this arm worked with a Community Health Worker (CHW) who provided a general health program that consisted of didactic information of unrelated general health information. Participants received the same number of contacts with their CHW as the intervention arm. Participants and CHW interacted by telephone 8 times over 3 months.
  Arms: General Health Program

SUMMARY:
As many as 75% of people with diabetes report chronic pain. While cognitive behavioral therapy (CBT) improves pain and functioning in individuals with chronic pain, many rural and underserved communities lack resources for such programs. The investigators tested the hypothesis that a CBT-based program delivered by community health workers (CHW) can improve quality of life in individuals with diabetes and chronic pain.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a growing chronic disease, affecting 20% of the population of Alabama. However, type 2 DM (90-95% of all DM) rarely occurs in isolation; 25% of all Americans report chronic pain, rising to 58-70% of community-dwellers over age 65. The National Center for Health Statistics reported in 2006 that chronic pain affected 76.2 million Americans, more than cancer, heart disease, stroke and DM combined. Despite the high prevalence of chronic pain, evidence suggests that under treatment is common. In one study, 68% of primary care physicians estimated that chronic pain was inadequately managed in their patients, and 60% thought improving physician education could help. Indeed, 40% of people with moderate to severe pain report not getting adequate relief.

Chronic pain is a significant barrier to successful DM self-care; patients with chronic pain have lower medication adherence and are less likely to exercise. Fully 60-80% of DM patients report chronic pain, and in our ENCOURAGE pilot study (Safford, PI), all but one participant did so. About 20-25% of pain may stem from neuropathy, but at least 1/3 stems from OA (osteoarthritis), and coexistence of multiple causes is common. Over half of patients >65 and 60% of women of any age report OA, demonstrating the very high prevalence of OA in this demographic group. Pain management dominated 20% of primary care visits for diabetic patients in one study, and decreased the likelihood of DM risk factor management. Not surprisingly, depressive symptoms are common in individuals with OA and chronic pain, and are also associated with non adherence to DM self-care behavior. Pain is therefore a barrier to not only quality of life, but to successful DM self-care.

While cognitive behavioral therapy (CBT) improves pain and functioning in individuals with chronic pain, many rural and underserved communities lack resources for such programs. The investigators tested the hypothesis that a CBT-based program delivered by community health workers (CHW) can improve quality of life in individuals with diabetes and chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* 19 or older in age
* diagnosed with diabetes
* under the care of a doctor
* experienced chronic pain in the past month

Exclusion Criteria:

* not community dwelling
* less than 19 years old
* pregnant
* end-stage medical conditions with limited life expectancy
* no access to telephone
* does not speak english,

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2011-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin (A1c) | change in A1c in 3 months
  fingerstick, point of care a1c test
Blood pressure | Change in blood pressure measure in 3 months
  measured using digital automated blood pressure monitor
Functional status (WOMAC) | change in functional status in 3 months
  Assessed using the the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Quality of Life (SF12) | Change in quality of life measures at 3 months
  self report using the Short form-12 (SF12)

SECONDARY OUTCOMES:
Pain (McGill Pain Questionnaire, ICOAP) | Change in pain measures at 3 months
  self report using the following measures: McGill Pain Questionnaire, A measure of intermittent and Constant Osteoarthritis Pain (ICOAP),
Body mass index (BMI) | change in BMI in 3 months
  weight measured using digital scale, height measured using stadiometer
Diabetes knowledge (Spoken Knowledge in Low Literacy in Diabetes Scale) | change in diabetes knowledge in 3 months
  assessed using a modified version of the Spoken Knowledge in Low Literacy in Diabetes Scale
diabetes management self-efficacy (PDSMS) | change in diabetes management self efficacy measures in 3 months
  assessed using the Perceived Diabetes Self-Management Scale (PDSMS)
Self efficacy in arthritis pain (Arthritis Self-Efficacy Scale) | change in pain self efficacy measures in 3 months
  assessed using the Pain Self Efficacy Subscale of the Arthritis Self-Efficacy Scale
Patient Activation Measure (PAM-13) | change in patient activation measures in 3 months
  assessed using the 13 item patient activation measure (PAM-13)
Perceived stress (PSS10) | change in perceived stress in 3 months
  Assessed using the Perceived Stress Scale (PSS10)
Pain coping strategies (CSQ24) | change in pain coping strategies in 3 months
  assessed using the pain coping strategies questionnaire (CSQ24)
Depressive symptoms (CESD-SF) | change in depressive symptoms in 3 months
  assessed using the Short Form of Center for Epidemiological Studies scale (CESD-SF)
Trust in physicians (Trust in Physicians Scale) | change in trust in physicians in 3 months
  assessed using the Trust in Physicians Scale
Medication Adherence (4-item Morisky Medication Adherence scale) | change in medication adherence in 3 months
  assessed using the 4-item Morisky Medication Adherence scale
Physical activity - usual daily activity | change in usual daily activity at 3 months
  participant self-report of usual daily activity (usually sit during the day, stand or walk but don't carry or lift things often, usually lift or carry light loads, or do heavy work or carry heavy loads)
Physical activity - number of days engaged in intense exercise in the past 7 days | change in days of intense exercise at 3 months
  participant self report of number of days in the past week engaged in intense exercise (0-7 days)
Physical activity - number of days walked for exercise in the past 7 days | change in days of walking for exercise at 3 months
  participant self report of number of days in the past week walked for exercise (0-7)
Physical activity - exercising when in pain questions | change exercising when in pain at 3 months
  participant self report of exercising when experiencing pain assessed by if the participant had no days unable to walk for exercise because of pain, unable to walk because of pain but did other exercises, or unable to walk because of pain but did not other forms of exercise.
Physical Activity - perception of physical activity compared to others | change in perception of physical activity at 3 months
  participant self report of activity levels compared to others their age
Diet - days eating high fat foods in the past 7 days | change in the number of days of eating high fat foods at 3 months
  participant self report of days in the past 7 days of eating high-fat foods
Diet - having a second serving at a meal in the past 7 days | change in the number of days of having a second serving at a meal in the past 7 days
  participant self report of days in the past 7 days of having a second serving at a meal in the past 7 days
Diet - eating unhealthy foods because of pain in the past 7 days | change in the number of days of eating unhealthy foods because of pain in the past 7 days at 3 months
  participant self report of days in the past 7 days of eating unhealthy foods because of experiencing pain

IPD SHARING:
Plan to Share IPD: No
The data will stay at UAB

REFERENCES:
- [Derived] Andreae SJ, Andreae LJ, Richman JS, Cherrington AL, Safford MM. Peer-delivered Cognitive Behavioral Therapy-based Intervention Reduced Depression and Stress in Community Dwelling Adults With Diabetes and Chronic Pain: A Cluster Randomized Trial. Ann Behav Med. 2021 Oct 4;55(10):970-980. doi: 10.1093/abm/kaab034. PMID 33969866
- [Derived] Andreae SJ, Andreae LJ, Richman JS, Cherrington AL, Safford MM. Peer-Delivered Cognitive Behavioral Training to Improve Functioning in Patients With Diabetes: A Cluster-Randomized Trial. Ann Fam Med. 2020 Jan;18(1):15-23. doi: 10.1370/afm.2469. PMID 31937528